CLINICAL TRIAL: NCT04761068
Title: Clinical Outcomes of Patients Undergoing Coronary Artery Bypass Grafting (CABG) Surgery With VEST Supported Venous Grafts
Brief Title: Clinical Outcomes of Patients Undergoing CABG Surgery With VEST Supported Venous Grafts
Status: Recruiting | Type: Observational
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Stefanos Demertzis, Head of cardiac surgery, Cardiocentro Ticino
Other Study IDs: VEST registry
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass surgery; CABG; External support
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: VEST — Venous External Support for vein grafts in CABG

SUMMARY:
This is a prospective, investigator-initiated, multi-center, open label and post-market registry, enrolling patients with atherosclerotic coronary artery disease, scheduled for CABG with at least one SVG bypass.

The registry is designed to evaluate the clinical outcome of CABG surgery with an external support device (VEST) for SVG bypasses.

In each patient, use of the VEST will be according to its approved indications for use and attempt will be made (based on clinical judgement) to support each non-sequential SVG bypass graft with a VEST device.

Subjects will be followed for 5 years, with interim follow ups at 12 and 24 months.

MACCE and EQ5D3L will be documented at every follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for planned CABG procedure with at least one SVG bypass with pre-planned VEST treatment.
2. Saphenous vein graft length and diameter are adequate for the planned intervention.
3. Patient is willing and able to give their written informed consent to participate in the registry study.
4. Patient is over 18 years of age

Exclusion Criteria:

1. Emergency CABG surgery (cardiogenic shock, inotropic pressure support, IABP)
2. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for planned CABG procedure with at least one SVG bypass with pre-planned VEST treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Ischemic driven target vessel revascularization | 5 years post Index CABG
  CABG or PCI of VEST supported vein graft or associated target coronary artery

SECONDARY OUTCOMES:
MACCE | 1, 2, and 5 years post index CABG
  The occurrence of any of the following major adverse cardiac and cerebrovascular events (MACCE): death; Stroke; Myocardial infarction (MI) and Coronary revascularization (redo-CABG and PCI).
Myocardial Infarction (MI) | 1, 2, and 5 years post index CABG
  Myocardial Infarction (MI)
Recurrent revascularization | 1, 2, and 5 years post index CABG
  Recurrent revascularization
Survival | 1, 2, and 5 years post index CABG
  Survival, both overall and freedom from cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Stefanos Demertzis, Principal Investigator — Cardiocentro Ticino
Locations (13):
- Austria (3):
  - Medical University of Innsbruck, Innsbruck
  - AKH (Vienna General Hospital), Vienna
  - Floridsdorf Clinic, Vienna
- Germany (3):
  - Herzzentrum Dresden, Dresden
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus der Barmherzigen Brüder, Trier
- Italy (2):
  - European hospital, Roma
  - Mauriziano Hospital, Turin
- Spain (3):
  - Germans Trias i Pujol, Badalona
  - University hospital of the Canary Islands, Santa Cruz de Tenerife
  - Ribera hospital, Valencia
- Switzerland (2):
  - Cardiocentro Ticino, Lugano
  - Triemli University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No